CLINICAL TRIAL: NCT02294331
Title: Attain Performa™ Left Ventricular Quadripolar Lead Post-Approval Study
Brief Title: Attain Performa™ Left Ventricular (LV) Quadripolar Leads Chronic Performance Study
Status: Completed | Type: Observational
Sponsor: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: Attain Performa™ PAS
Record Dates: First submitted 2014-10-08; First posted 2014-11-19 (Estimated); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Attain Performa™ LV Leads: Patients who meet all Inclusion criteria and no Exclusion criteria and are implanted with an Attain Performa™ LV lead.

SUMMARY:
Lead survivability will be summarized.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate long-term performance of the Attain Performa™ LV Leads. This evaluation is based on the number of lead-related complications occurring during the study compared to the number of leads enrolled in the study. The leads will be followed for 5 years after implant. This study is required by FDA as a condition of approval of the Attain Performa™ LV Leads. This study is conducted within Medtronic's post-market surveillance platform.

ELIGIBILITY:
Patients who meet all of the following inclusion criteria and do not meet any of the following exclusion criteria are eligible for enrollment.

Inclusion Criteria

* Patient or legally authorized representative provides written authorization and/or consent per institution and geographical requirements
* Patient has or is intended to receive an Attain Performa™ LV lead
* Patient within 30 day post implant enrollment window

Exclusion Criteria

* Patient who is, or is expected to be inaccessible for follow-up
* Patient with exclusion criteria required by local law
* Patient is currently enrolled in or plans to enroll in any concurrent drug and/or device study that may confound results

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients implanted with an Attain Performa™ LV Lead within 30 days. All subjects must meet Inclusion criteria and none of the Exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1900 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Lead complication | 5 years
  Survival analysis will be used to analyze the lead. Lead status will be reported as a function of time post-implant for all leads in the study.
  Lead related complications include but are not limited to: failure to capture, abnormal sensing, threshold rise, abnormal impedance, insulation breach, conductor fracture, extracardiac stimulation, lead dislodgement, cardiac perforation, structural lead failure.

SECONDARY OUTCOMES:
Types of lead-related adverse device effects | 5 years
  Summary statistics will be used to report types and rates of lead related adverse device effects (ADE). Examples of ADEs include but are not limited to: failure to capture, abnormal sensing, threshold rise, abnormal impedance, insulation breach, conductor fracture, extracardiac stimulation, lead dislodgement, cardiac perforation, structural lead failure.
Returned lead analysis | 5 years
  A listing of analysis results of all Attain Performa study leads which are explanted and returned for analysis will be reported.
Lead survival estimate by model | 5 years
  An analysis will be conducted at the end of the study to provide comparative statistics on the safety performance of each individual lead model.

CONTACTS AND LOCATIONS:
Locations (100):
- United States (81):
  - Birmingham, Alabama
  - Anchorage, Alaska
  - Chandler, Arizona
  - Gilbert, Arizona
  - Jonesboro, Arkansas
  - Bakersfield, California
  - Rancho Mirage, California
  - Redwood City, California
  - Salinas, California
  - San Diego, California
  - Stanford, California
  - Torrance, California
  - Van Nuys, California
  - Colorado Springs, Colorado
  - Lakewood, Colorado
  - New Haven, Connecticut
  - Washington D.C., District of Columbia
  - Bradenton, Florida
  - Clearwater, Florida
  - Jacksonville, Florida
  - Safety Harbor, Florida
  - Albany, Georgia
  - Marietta, Georgia
  - Evansville, Indiana
  - West Des Moines, Iowa
  - Kansas City, Kansas
  - Edgewood, Kentucky
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Baton Rouge, Louisiana
  - Hyattsville, Maryland
  - Salisbury, Maryland
  - Silver Spring, Maryland
  - Takoma Park, Maryland
  - Lansing, Michigan
  - Marquette, Michigan
  - Ypsilanti, Michigan
  - Minneapolis, Minnesota
  - Robbinsdale, Minnesota
  - Rochester, Minnesota
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Columbia, Missouri
  - Kansas City, Missouri
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Lebanon, New Hampshire
  - Morristown, New Jersey
  - Albuquerque, New Mexico
  - Huntington, New York
  - New York, New York
  - Poughkeepsie, New York
  - Utica, New York
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Raleigh, North Carolina
  - Akron, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Toledo, Ohio
  - Portland, Oregon
  - Allentown, Pennsylvania
  - St Luke's University Health Network, Bethlehem, Pennsylvania
  - Danville, Pennsylvania
  - Erie, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Wilkes-Barre, Pennsylvania
  - Germantown, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Plano, Texas
  - The Woodlands, Texas
  - Burlington, Vermont
  - Falls Church, Virginia
  - Leesburg, Virginia
  - Spokane, Washington
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
- Leuven, Belgium
- Canada (6):
  - Calgary, Alberta
  - London, Ontario
  - Montreal, Quebec
  - Québec, Quebec
  - Calgary
  - Ottawa
- France (2):
  - La Rochelle
  - Nantes
- Germany (3):
  - Essen
  - Hanover
  - Ulm
- Netherlands (4):
  - Eindhoven
  - Maastricht
  - Nieuwegein
  - Rotterdam
- Zurich, Switzerland
- United Kingdom (2):
  - Liverpool
  - Middlesbrough